CLINICAL TRIAL: NCT04101656
Title: Accelerated Partial Irradiation of the Breast: New Altered Fractionation
Status: Recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-APBI-2019-02
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Radiotherapy; Accelerated Partial Breast Irradiation; APBI; Modulated Intensity Radiotherapy; IMRT; Positive estrogen receptor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: APBI (Accelerated Partial Breast Irradiation): APBI 28 Gy in 5 fractions of 5.6 Gy, using external radiotherapy with modulated intensity technique (IMRT)

SUMMARY:
The aim of this observational study is to evaluate a dose fractionation scheme for APBI using external radiotherapy with modulated intensity technique (IMRT), with the possible impact on the quality of life of patients as it decreases the treatment number of sessions and improves the efficiency and accessibility.

DETAILED DESCRIPTION:
Breast cancer is the most common tumor among women; although its treatment used to be very aggressive, nowadays is based on the minimum effective treatment.

In non-metastatic patients, the therapeutical strategy is based on surgery, systemic therapy and radiotherapy. Usually in the early stages of the disease, the treatment begins with a conservative surgery followed by adjuvant therapy.

It´s been proved that the majority of relapses after conservatory surgery occur near the surgical bed which suggests that the main benefit of radiotherapy treatment lies in its primary effect on residual microscopic disease in the surgical bed. Regarding the radiotherapy used after conservative surgery, it´s accepted as standard treatment hypofractionated schemes, after they have demonstrated at least the same grade of effectiveness as the classic fractionation in terms of locoregional control, survival, aesthetic results or toxicity.

One of the options of hypofractionated schemes is APBI (Accelerated Partial Breast Irradiation), that by reducing the volume of the radiated breast and an accelerated dose fractionation scheme, can eliminate the residual microscopic disease in the surgical bed. The main advantage of APBI is that can shorten the overall time (total treatment time) by increasing the dose per fraction.

In patients who meet the following criteria:≥ 45 years or 40-44 if there isn´t any other risk factor, diagnosed with infiltrating ductal carcinoma (IDC) or ductal carcinoma in situ (DCIS) and that have undergone conservative surgery without ganglionar involvement (pN0) of any histological degree except from invasive lobular carcinoma and with a size ≤ 3 cm, with a free margin of at least 2 mm, as well as with positive and negative estrogen receptor tumors; APBI is currently considered standard treatment.

This radiotherapy modality can be administered using 4 different techniques: interstitial brachytherapy, spherical balloons, intraoperative radiotherapy with electrons or with dedicated kilovoltage (RIO) systems and External Radiotherapy (3D shaped RT or modulated intensity radiotherapy - IMRT-). Each of them have their advantages and disadvantages, without any of them being superior to the others in terms of survival or local control, however, IMRT achieves a more shaped and uniformed dose after conservative surgery.

The aim of this observational study is to evaluate a dose fractionation scheme for APBI (28 Gy in 5 fractions of 5.6 GY, 5 days/week) using external radiotherapy with modulated intensity technique (IMRT), with the possible impact on the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 45 years or 40-44 if there isn´t any other risk factor
* Diagnosed with infiltrating ductal carcinoma (IDC) or ductal carcinoma in situ (DCIS) and that have undergone conservative surgery without ganglionar involvement (pN0) of any histological degree except from invasive lobular carcinoma and with a size ≤ 3 cm.
* Disease free margins (R0: > 2mm).
* Positive and negative estrogen receptor tumors.

Exclusion Criteria:

* Multicentric and multifocal tumors, except from if it´s focal and the only risk factor.
* Patients must not have undergone a neoadjuvant QT therapy.
* Patients with BRCA positive mutation will be excluded.
* Those patients unable or unsuitable to understand and accept the informed consent.
* Metastasic´s affectation evidence.
* Extensive lymphovascular invasion, except from if the total resulting size of the focus and breast parenchyma addition is ≤ 3cm.
* Breast implants presence in the breast that´s going to be treated.
* Contraindicated radiotherapy treatment due to a diagnosis of cutaneous lupus, pregnancy or scleroderma.
* Inability to fully know the dosimetric data of the APBI plan.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients that meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the security in terms of acute toxicity | Up to 5 years after the end of the irradiation
  Adverse effects due to radiotherapy

SECONDARY OUTCOMES:
Dose analysis in critical organs | Up to 5 years after the end of the irradiation
  Measurement of dose in the heart, ipsilateral and contralateral lung, ipsilateral and contralateral breast taking into account the acceptable and optimal dose limit.
Evaluate chronic toxicity | Up to 5 years after the end of the irradiation
  Adverse effects due to radiotherapy
Verify the incidence of locoregional tumor relapses at 2 and 5 years of follow-up | Up to 5 years after the end of the irradiation
  Clinical or imaged based detection of the already treated breast cancer tumor (local relapse) or the ipsilateral regional ganglionic chains: armpit, supraclavicular cavity or internal breast chain (regional relapse).
Verify the disease free survival at 2 and 5 years of follow-up | Up to 5 years after the end of the irradiation
  The disease free survival is the time that passes from the end of the treatment until a control is done or takes place a relapse (local or distant).
Verify the disease overall survival at 2 and 5 years of follow-up | Up to 5 years after the end of the irradiation
  The disease overall survival is the time that passes from the end of the treatment until a control is done or the patient´s death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain